CLINICAL TRIAL: NCT03808285
Title: Denosumab Related Osteonecrossi of the Jaw : : an Emergent and Potentially Complex Bone and Joint Infection
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Eugénie MABRUT, Clinical Research Assistant, Hospices Civils de Lyon
Other Study IDs: 18-334
Record Dates: First submitted 2019-01-04; First posted 2019-01-17 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Bone and Joint Infection; Osteomyelitis; Adverse Drug Event
Keywords: bone and joint infection; osteomyelitis; mandibular; denosumab
MeSH Terms: conditions — Osteomyelitis; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mandibular osteomylitis: description of mandibular osteomylitis due to denosumab
  Interventions: Other: mandibular osteomylitis

INTERVENTIONS:
Other: mandibular osteomylitis

SUMMARY:
The aim of this study is to adescription of mandibular osteomylitis in patients having had a treatment by DENOSUMAB. Indeed, one of the adverse effect ot this molecule is to induce mandibular infection.

ELIGIBILITY:
Inclusion Criteria:

* patients having a mandibular osteomylelitis due to DENOSUMAB

Exclusion Criteria:

* none

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients having a mandibular osteomylelitis due to DENOSUMAB betwwen 01/01/2013 and 31/12/2018 and managed at the Lyon Bone and joint infection refence Center
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of mandibular osteomyelitis | Entire description can be made at the outcome which is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  description of mandibular osteomyelitis

SECONDARY OUTCOMES:
Duration of antibiotics | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  Description of the duration and strategies of antibiotic treatments used (double-agent therapy, monotherapy)
Rate of Treatment Failure | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin. Analyse of risk factor.
management of mandibular osteomyelitis by medical team | all data are available at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  description of medical and surgical strategies : data availables in consultation report

CONTACTS AND LOCATIONS:
Overall Officials: TRISTAN FERRY, MD,PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided